CLINICAL TRIAL: NCT03776812
Title: A Phase 2, Randomized, Open-Label, 3-arm Study of Relacorilant in Combination With Nab-Paclitaxel for Patients With Recurrent Platinum-Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Study of Relacorilant in Combination With Nab-Paclitaxel for Patients With Recurrent Platinum-Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORT125134-552
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Ovarian Cancer; Recurrent Fallopian Tube Carcinoma; Recurrent Primary Peritoneal Carcinoma
Keywords: Glucocorticoid Receptor; Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; Nab-paclitaxel; Glucocorticoid Receptor Antagonist; Relacorilant
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — relacorilant; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Continuous Relacorilant Dosing (Experimental): Patients will receive relacorilant 100 mg (titrated up to 150 mg after Cycle 1 or 2) once daily in combination with nab-paclitaxel 80 mg/m^2, on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: Relacorilant; Drug: Nab-paclitaxel
- Arm B: Intermittent Relacorilant Dosing (Experimental): Patients will receive relacorilant 150 mg on the day before (excluding Cycle 1, Day -1), the day of, and the day after nab-paclitaxel, in combination with nab-paclitaxel 80 mg/m^2, on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: Relacorilant; Drug: Nab-paclitaxel
- Arm C: Nab-paclitaxel Comparator (Active Comparator): Patients will receive nab-paclitaxel 100 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle. Patients initially in Arm C who choose to cross over after disease progression will receive relacorilant 100 mg (titrated up to 150 mg) in combination with nab-paclitaxel 80 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle after cross over.
  Interventions: Drug: Relacorilant; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Relacorilant — Relacorilant is supplied as capsules for oral dosing.
Drug: Nab-paclitaxel — Nab-paclitaxel is administered as IV infusion over 30-40 minutes.
  Other Names: Abraxane

SUMMARY:
This is a Phase 2, open-label, randomized, 3-arm study to evaluate progression-free survival (PFS) in patients with recurrent platinum-resistant ovarian, fallopian tube, or primary peritoneal cancer treated with intermittent or continuous regimens of relacorilant in combination with nab-paclitaxel compared with patients treated with nab-paclitaxel alone.

DETAILED DESCRIPTION:
Relacorilant is a small molecule antagonist of the glucocorticoid receptor (GR). The goals of this study are to evaluate the efficacy of relacorilant either administered daily (continuous) or on the day prior, the day of, and the day after chemotherapy (intermittent) in combination with nab-paclitaxel in the treatment of platinum-resistant ovarian, fallopian tube, or primary peritoneal cancers compared with nab-paclitaxel alone. The safety, pharmacokinetics (PK), and pharmacodynamic profile of relacorilant in combination with nab-paclitaxel will also be assessed.

Eligible patients will be randomized 1:1:1 to one of the following three treatment arms. Patient randomization will be stratified by treatment-free interval from most recent taxane (relapsed within 6 months vs >6 months) and presence of ascites (yes vs no).

* Arm A (Continuous relacorilant): Relacorilant starting at 100 mg, administered orally, once daily every day in combination with nab-paclitaxel on Days 1, 8, and 15 of each 28-day cycle.
* Arm B (Intermittent relacorilant): Relacorilant 150 mg, administered orally, on the day before (excluding Cycle 1, Day -1), the day of, and the day after nab-paclitaxel, in combination with nab-paclitaxel on Days 1, 8, and 15 of each 28-day cycle.
* Arm C (Comparator): Nab-paclitaxel on Days 1, 8, and 15 of each 28-day cycle.

Patients will remain on study treatment until reaching a protocol-defined event of disease progression (PD), experiencing unmanageable toxicity, or until other treatment discontinuation criteria are met. All patients will be followed for progression, subsequent therapies, and survival in the long-term follow-up phase. Patients in Arm C who experience unequivocal PD per RECIST v1.1 will be given the opportunity to receive relacorilant in combination with nab-paclitaxel after discussion with the Medical Monitor (Crossover patients).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Investigational Review Board/Independent Ethics Committee-approved informed consent form (ICF) prior to study-specific screening procedures.
* Female patients aged ≥18 years old at time of consent
* Histologic diagnosis of high grade serous or endometrioid epithelial ovarian, primary peritoneal, or fallopian tube cancer or ovarian carcinosarcoma. Clear cell, mucinous and borderline histologic subtypes are excluded.
* Received at least 1 line of therapy with evidence of cancer progression within 6 months after the last dose of platinum-based therapy (ie, having a platinum-free interval of ≤6 months [platinum resistant]), or progressive disease during or immediately after primary platinum-therapy, (ie, platinum refractory). Patients with primary platinum resistance (progression within 6 months of the last dose of first-line platinum-containing chemotherapy) are considered eligible.

Notes: For the calculation of the platinum-free interval, cancer progression must be defined by clear evidence of progression, such as radiographic progression per RECIST v1.1. Calculating the platinum-free interval on the basis of increased Cancer Antigen (CA-125) is not allowed.

* Measurable or non-measurable disease by RECIST v1.1:

  * Previously irradiated lesions are not allowed as measurable disease, unless there is documented evidence of progression in the lesions.
  * To be eligible with non-measurable disease, patients must have evaluable disease with CA 125 at least twice the upper limit of reference range (of CA-125 ≥70 U/mL), along with radiographically evaluable disease by computerized tomography (CT)/magnetic resonance imaging (MRI).
* Availability and consent to provide tumor tissue for biomarker assays (archival or recent biopsy).
* No more than 4 prior chemotherapeutic or myelosuppressive regimens (not including maintenance therapy such as single-agent bevacizumab or poly (ADP-ribose) polymerase [PARP] inhibitors). Patients with platinum-refractory cancer cannot have had more than 2 prior lines of treatment for refractory disease.
* Appropriate to treat with nab-paclitaxel, in the opinion of the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Adequate organ and bone marrow function meeting the following criteria at the Screening Visit:

  * Absolute neutrophil count (ANC) ≥1,500 cells/mm^3.
  * Platelet count ≥100,000/mm^3.
  * Hemoglobin ≥9 g/dL.
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN) (or ≤5 × ULN in the context of liver metastasis).
  * Total bilirubin ≤1.5 × ULN.
  * Creatinine clearance ≥45 mL/min/1.73 m^2 (measured or estimated).
  * Albumin ≥3 g/dL (≥30 g/L) .
* If patient has undergone surgery of the gastrointestinal or hepatobiliary tract, adequate absorption as evidenced by: albumin ≥3.0 g/dL, controlled pancreatic insufficiency (if present), and lack of malabsorption.
* Able to swallow and retain oral medication and does not have uncontrolled emesis.
* Able to comply with protocol requirements.
* Negative pregnancy test for patients of childbearing potential. Patients of childbearing potential must use appropriate precautions to avoid pregnancy, defined as of non-childbearing potential (ie, postmenopausal or permanently sterilized) or using highly effective contraception with low user-dependency, for at least 3 months after the last dose of relacorilant, or per the duration indicated in the product label for nab-paclitaxel, whichever is latest. A woman is postmenopausal if it is more than 12 months since her last menstruation, without an alternative medical cause. Accepted methods of permanent sterilization methods are hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy. Accepted methods of highly effective contraception with low-user-dependency are:

  * An intrauterine device (IUD), provided that the subject has tolerated its use for at least 3 months before the first dose of study medication and undertakes not to have it removed for 1 month after the last dose.
  * Abstinence from heterosexual intercourse, when it is in line with the subject's preferred and usual lifestyle. Periodic abstinence and withdrawal are NOT acceptable.
  * Vasectomized partner provided that the partner is the sole sexual partner of the trial participant and that the vasectomized partner has received medical assessment of the surgical success.
  * Oral hormonal contraceptives are NOT permitted.

Exclusion Criteria:

* Clinically relevant toxicity from prior systemic anticancer therapies or radiotherapy that in the opinion of the Investigator has not resolved to Grade 1 or less prior to randomization.
* Any major surgery within 4 weeks prior to randomization. If subject received major surgery including (curative or palliative surgery), they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Treatment with the following prior to randomization:

  * Concurrent treatment with other anticancer therapy including other chemotherapy, immunotherapy, radiotherapy, chemoembolization, targeted therapy, an investigational agent or the non-approved use of a drug or device within 28 days before the first dose of study drug.
  * Hormonal anticancer therapies within 7 days of the first dose of study drug.
  * Systemic, inhaled, or prescription strength topical corticosteroids within 21 days of the first dose of study drug. Short courses (≤5 days) for non-cancer-related reasons are allowed if clinically required (such as prophylaxis for CT).
* Received radiation to more than 25% of marrow-bearing areas.
* Toxicities of prior therapies (except alopecia) that have not resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 ≤Grade 1.
* Requirement for treatment with chronic or frequently used oral corticosteroids for medical conditions or illnesses (eg, rheumatoid arthritis, immunosuppression after organ transplantation).
* History of severe hypersensitivity or severe reaction to either study drug.
* Peripheral neuropathy from any cause >Grade 1.
* Pregnant or lactating patients or patients expecting to conceive children within the projected duration of the trial, starting with the Screening Visit through at least 3 months after the last dose of relacorilant, or per the duration indicated in the product label for nab-paclitaxel, whichever is latest.
* Human immunodeficiency virus or current chronic/active infection with hepatitis C virus or hepatitis B virus, including:

  * Patients with chronic or active hepatitis B as diagnosed by serologic tests are excluded from the study. In equivocal cases, hepatitis B or C polymerase chain reaction may be performed and must be negative for enrollment.
* Patient has a clinically significant uncontrolled condition(s) or which in the opinion of the Investigator may confound the results of the trial or interfere with the patient's participation, including but not limited to:

  * Unstable angina pectoris, angioplasty, cardiac stenting, or myocardial infarction 6 months before study entry.
  * Uncontrolled hypertension (sustained systolic blood pressure >150 mmHg or diastolic pressure >100 mmHg despite optimal management). Patients will be considered eligible if hypertension is treated and controlled during Screening.
  * Active infection that requires parenteral antibiotics.
  * Bowel obstruction or gastric outlet obstruction.
  * Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Untreated parenchymal central nervous system metastases.
* Any other concurrent cancer or a history of another invasive malignancy within the last 3 years that has a likelihood of recurrence of >30% within the next 5 years. Adequately treated non-melanoma skin cancers or non-muscle invasive urothelial cancer or other tumors curatively treated with no evidence of disease are permissible.
* Are taking a concomitant medication that is a strong CYP3A inhibitor or inducer, or that is a substrate of CYP3A with a narrow therapeutic window.
* Concurrent treatment with mifepristone or other glucocorticoid receptor (GR) antagonists.
* Concurrent treatment on other investigational treatment studies for the treatment of ovarian, fallopian tube, or primary peritoneal cancer.
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only patients with recurrent ovarian, primary peritoneal, or fallopian tube cancer will be considered for this study
Enrollment: 178 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Pai, MD, Study Director — Corcept Therapeutics
Locations (24):
- United States (12):
  - Site Reference ID/Investigator #004, Birmingham, Alabama
  - Site Reference ID/Investigator #038, Scottsdale, Arizona
  - Site Reference ID/Investigator #032, Denver, Colorado
  - Site Reference ID/Investigator #001, Chicago, Illinois
  - Site Reference ID/Investigator #106, Boston, Massachusetts
  - Site Reference ID/Investigator #128, Boston, Massachusetts
  - Site Reference ID/Investigator #051, New York, New York
  - Site Reference ID/Investigator #169, New York, New York
  - Site Reference ID/Investigator #170, New York, New York
  - Site Reference ID/Investigator #127, Pittsburgh, Pennsylvania
  - Site Reference ID/Investigator #135, Charlottesville, Virginia
  - Site Reference ID/Investigator #121, Milwaukee, Wisconsin
- Belgium (3):
  - Site Reference ID/Investigator #109, Brussels
  - Site Reference ID/Investigator #119, Edegem
  - Site Reference ID/Investigator #108, Leuven
- Canada (2):
  - Site Reference ID/Investigator #117, Toronto, Ontario
  - Site Reference ID/Investigator #096, Montreal, Quebec
- Italy (3):
  - Site Reference ID/Investigator #122, Milan
  - Site Reference ID/Investigator #112, Napoli
  - Site Reference ID/Investigator #124, Roma
- Spain (4):
  - Site Reference ID/Investigator #115, Barcelona
  - Site Reference ID/Investigator #114, Madrid
  - Site Reference ID/Investigator #116, Madrid
  - Site Reference ID/Investigator #113, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou Y, Tong F, Jin B, Pan J, Ren N, Ren L, Xu Q. Relacorilant plus nab-paclitaxel for recurrent, platinum-resistant ovarian cancer: a cost-effectiveness study. J Gynecol Oncol. 2025 Jul;36(4):e63. doi: 10.3802/jgo.2025.36.e63. Epub 2025 Feb 20. PMID 40051286
- [Derived] Colombo N, Van Gorp T, Matulonis UA, Oaknin A, Grisham RN, Fleming GF, Olawaiye AB, Nguyen DD, Greenstein AE, Custodio JM, Pashova HI, Tudor IC, Lorusso D. Relacorilant + Nab-Paclitaxel in Patients With Recurrent, Platinum-Resistant Ovarian Cancer: A Three-Arm, Randomized, Controlled, Open-Label Phase II Study. J Clin Oncol. 2023 Oct 20;41(30):4779-4789. doi: 10.1200/JCO.22.02624. Epub 2023 Jun 26. PMID 37364223

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The intent-to-treat (ITT) population included all randomized patients.
Period: Overall Study
Arm/Group | Arm A: Continuous Relacorilant Dosing | Arm B: Intermittent Relacorilant Dosing | Arm C: Nab-paclitaxel Comparator
Started | 58 | 60 | 60
Entered Crossover | 0 | 0 | 28
Completed | 0 | 0 | 0
Not Completed | 58 | 60 | 60
Not completed — Death | 53 | 49 | 56
Not completed — Withdrawal by Subject | 1 | 7 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Did not enter long-term follow-up | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Population: The ITT population included all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Continuous Relacorilant Dosing | Arm B: Intermittent Relacorilant Dosing | Arm C: Nab-paclitaxel Comparator | Total
Number analyzed (Participants) | 58 | 60 | 60 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (8.8) | 60.3 (9.7) | 61.8 (8.8) | 60.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 60 | 60 | 178
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6 | 12
  Not Hispanic or Latino | 53 | 54 | 49 | 156
  Unknown or Not Reported | 2 | 3 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 1 | 2
  White | 57 | 52 | 50 | 159
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: To assess time from randomization until the date of first documented progressive disease (PD) by RECIST v1.1 (as determined by the Investigator at the local site), or death due to any cause, whichever occurs first.
Time Frame: Baseline and up to 15 months
Population: The ITT population included all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Continuous Relacorilant Dosing | Arm B: Intermittent Relacorilant Dosing | Arm C: Nab-paclitaxel Comparator
Number analyzed (Participants) | 58 | 60 | 60
months | 5.29 [3.84 to 5.55] | 5.55 [3.68 to 7.20] | 3.76 [3.52 to 5.36]
Statistical Analysis 1: Comparison: Arm A: Continuous Relacorilant Dosing vs Arm C: Nab-paclitaxel Comparator; Test type: Other; p = 0.3293, Cox proportional hazards model; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.56 to 1.22]
Statistical Analysis 2: Comparison: Arm B: Intermittent Relacorilant Dosing vs Arm C: Nab-paclitaxel Comparator; Test type: Other; p = 0.0384, Cox proportional hazards model; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.44 to 0.98]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: To assess the proportion of patients with measurable disease at Baseline who attain complete response (CR) or partial response (PR) by RECIST v1.1 (confirmation not required).
Time Frame: Baseline and up to 15 months
Population: Patients in the ITT population with measurable disease at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Continuous Relacorilant Dosing | Arm B: Intermittent Relacorilant Dosing | Arm C: Nab-paclitaxel Comparator
Number analyzed (Participants) | 54 | 56 | 53
Participants | 19 | 20 | 19

3. Secondary Outcome: Duration of Response (DOR)
Description: To assess the time from when response (CR or PR) was first documented to the first objectively documented PD or death (whichever occurs first)
Time Frame: From first documented response up to 12 months
Population: Patients in the ITT population with measurable disease at Baseline and who attain CR or PR by RECIST v1.1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Continuous Relacorilant Dosing | Arm B: Intermittent Relacorilant Dosing | Arm C: Nab-paclitaxel Comparator
Number analyzed (Participants) | 19 | 20 | 19
months | 3.79 [2.33 to 5.55] | 5.55 [3.75 to 5.88] | 3.65 [2.89 to 5.09]

4. Secondary Outcome: Cancer Antigen 125 (CA-125) Response According to Gynecological Cancer Intergroup Criteria (GCIG)
Description: To assess the overall CA-125 response per GCIG criteria. Response was defined as ≥50% reduction in CA-125 from a pre-treatment sample. Patients whose CA-125 levels fall within the reference range are classified as complete responders.
Time Frame: Baseline and up to 15 months
Population: Patients in the ITT population with an initial CA-125 level ≥ twice the upper limit of normal (ULN) of the reference range.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Continuous Relacorilant Dosing | Arm B: Intermittent Relacorilant Dosing | Arm C: Nab-paclitaxel Comparator
Number analyzed (Participants) | 51 | 53 | 52
Participants | 32 | 34 | 28

5. Secondary Outcome: Best Overall Response (BOR)
Description: To assess the best response (CR, PR, stable disease [SD], or PD) recorded from the date of randomization until PD/recurrence (or death)
Time Frame: Baseline and up to 15 months
Population: Patients in the ITT population with measurable disease at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Continuous Relacorilant Dosing | Arm B: Intermittent Relacorilant Dosing | Arm C: Nab-paclitaxel Comparator
Number analyzed (Participants) | 54 | 56 | 53
Participants
  Complete response | 4 | 1 | 2
  Partial response | 15 | 19 | 17
  Stable disease | 23 | 20 | 21
  Progressive disease | 9 | 14 | 12
  Not evaluable | 3 | 2 | 1

6. Secondary Outcome: PFS Rate at 6 and 12 Months
Description: To assess the proportion of patients who have not progressed according to RECIST v1.1 criteria at 6 and 12 months. Values are Kaplan-Meier estimates of the patients progression-free at the time points specified.
Time Frame: 6 and 12 months
Population: The ITT population included all randomized patients.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Arm A: Continuous Relacorilant Dosing | Arm B: Intermittent Relacorilant Dosing | Arm C: Nab-paclitaxel Comparator
Number analyzed (Participants) | 58 | 60 | 60
proportion of patients
  6 months | 0.26 [0.15 to 0.38] | 0.40 [0.28 to 0.53] | 0.25 [0.15 to 0.36]
  12 months | 0.08 [0.02 to 0.18] | 0.11 [0.04 to 0.23] | 0.04 [0.01 to 0.12]

7. Secondary Outcome: PFS in Patients Who Cross Over to Continuous Treatment at Time of Initial PD
Description: To assess the time from crossover Baseline (initial PD) until the earliest date of subsequent PD by RECIST v1.1, as determined by the Investigator at the local site, or death from any cause, whichever comes first.
Time Frame: Crossover Baseline (Day 50) up to Day 272
Population: Patients in the ITT population initially in Arm C: Nab-paclitaxel Comparator, who choose to cross over after disease progression.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Crossover Patients: Patients initially in the Nab-paclitaxel Comparator Arm C who choose to cross over after disease progression will receive relacorilant 100 mg (titrated up to 150 mg) in combination with nab-paclitaxel 80 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle after cross over.
Arm/Group | Crossover Patients
Number analyzed (Participants) | 27
months | 2.10 [1.87 to 2.50]

8. Secondary Outcome: ORR in Patients Who Cross Over to Continuous Treatment at Time of Initial PD
Description: To assess the proportion of patients with measurable disease at the crossover Baseline who attain confirmed CR or PR by RECIST v1.1
Time Frame: Crossover Baseline (Day 50) up to Day 272
Population: Patients in the ITT population initially in Arm C: Nab-paclitaxel Comparator, who choose to cross over after disease progression and have measurable disease at the crossover Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Crossover Patients
Number analyzed (Participants) | 21
Participants | 0

9. Secondary Outcome: DOR in Patients Who Cross Over to Continuous Treatment at Time of Initial PD
Description: To assess the time from when the first objective response (CR or PR) in the crossover period to the first objectively documented subsequent PD, or death (whichever occurs first)
Time Frame: From the time of objective response in the crossover period to the time of subsequent PD
Population: No crossover patients attained CR or PR, so duration of response could not be analyzed.
Arm/Group | Crossover Patients
Number analyzed (Participants) | 0

10. Secondary Outcome: BOR in Patients Who Cross Over to Continuous Treatment at Time of Initial PD
Description: To assess the best overall response (CR, PR, SD, or PD) recorded in the crossover period
Time Frame: Crossover Baseline (Day 50) up to Day 272
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Crossover Patients
Number analyzed (Participants) | 21
Participants
  Complete response | 0
  Partial response | 0
  Stable disease | 3
  Progressive disease | 18
  Not evaluable | 0

11. Secondary Outcome: Overall Survival (OS)
Description: To assess the time from randomization to death by any cause.
Time Frame: Up to 31 months
Population: The ITT population included all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Continuous Relacorilant Dosing | Arm B: Intermittent Relacorilant Dosing | Arm C: Nab-paclitaxel Comparator
Number analyzed (Participants) | 58 | 60 | 60
months | 11.30 [7.52 to 16.39] | 13.90 [11.07 to 18.43] | 12.19 [7.72 to 15.28]

12. Secondary Outcome: Overall Response According to Combined RECIST v1.1 + GCIG Criteria
Description: To assess the proportion of patients with measurable disease at Baseline who attain confirmed CR or PR by RECIST v1.1 and GCIG criteria. GCIG response was defined as ≥50% reduction in CA-125 from a pre-treatment sample.
Time Frame: Baseline and up to 15 months
Population: Patients in the ITT population with an initial CA-125 level ≥ twice the ULN of the reference range within 2 weeks before starting treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Continuous Relacorilant Dosing | Arm B: Intermittent Relacorilant Dosing | Arm C: Nab-paclitaxel Comparator
Number analyzed (Participants) | 58 | 60 | 60
Participants | 34 | 36 | 33

ADVERSE EVENTS:
Time Frame: Up to 39 months
Description: All-Cause Mortality: the ITT population. Serious Adverse Events and Other (not including serious) Adverse Events: the safety population included all randomized patients who received ≥1 dose of study treatment.
Arm/Group | Arm A: Continuous Relacorilant Dosing | Arm B: Intermittent Relacorilant Dosing | Arm C: Nab-paclitaxel Comparator
All-Cause Mortality (participants affected / at risk) | 53/58 | 49/60 | 56/60
Serious Adverse Events (participants affected / at risk) | 30/57 | 15/60 | 19/60
Other Adverse Events (participants affected / at risk) | 57/57 | 59/60 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Continuous Relacorilant Dosing (N=57) | Arm B: Intermittent Relacorilant Dosing (N=60) | Arm C: Nab-paclitaxel Comparator (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 5 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Biliary tract infection (Infections and infestations) | 0 | 0 | 1
Coronavirus infection (Infections and infestations) | 0 | 1 | 0
Escherichia pyelonephritis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0
Stoma site abscess (Infections and infestations) | 0 | 0 | 1
Subperiosteal abscess (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Malignant ascites (Gastrointestinal disorders) | 1 | 2 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0
Paraneoplastic neurological syndrome (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Pleural efffusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Melanocytic hyperplasia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Bacterial diarrhoea (Infections and infestations) | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Stoma prolapse (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Continuous Relacorilant Dosing (N=57) | Arm B: Intermittent Relacorilant Dosing (N=60) | Arm C: Nab-paclitaxel Comparator (N=60)
Anaemia (Blood and lymphatic system disorders) | 39 | 29 | 34
Neutropenia (Blood and lymphatic system disorders) | 20 | 11 | 20
Leukopenia (Blood and lymphatic system disorders) | 7 | 3 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 2 | 5
Tachycardia (Cardiac disorders) | 5 | 1 | 1
Palpitations (Cardiac disorders) | 4 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 3 | 1
Lacrimation increased (Eye disorders) | 8 | 6 | 2
Visual impairment (Eye disorders) | 4 | 0 | 3
Dry eye (Eye disorders) | 2 | 3 | 1
Nausea (Gastrointestinal disorders) | 41 | 30 | 27
Constipation (Gastrointestinal disorders) | 25 | 19 | 17
Abdominal pain (Gastrointestinal disorders) | 21 | 16 | 20
Vomiting (Gastrointestinal disorders) | 27 | 18 | 15
Diarrhoea (Gastrointestinal disorders) | 22 | 16 | 15
Abdominal pain upper (Gastrointestinal disorders) | 7 | 9 | 6
Stomatitis (Gastrointestinal disorders) | 15 | 3 | 3
Abdominal distension (Gastrointestinal disorders) | 9 | 6 | 4
Dyspepsia (Gastrointestinal disorders) | 7 | 4 | 4
Ascites (Gastrointestinal disorders) | 6 | 5 | 4
Abdominal discomfort (Gastrointestinal disorders) | 3 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 4
Fatigue (General disorders) | 19 | 19 | 21
Asthenia (General disorders) | 24 | 15 | 19
Oedema peripheral (General disorders) | 8 | 10 | 12
Pyrexia (General disorders) | 5 | 6 | 10
Peripheral swelling (General disorders) | 4 | 3 | 3
Malaise (General disorders) | 5 | 1 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 3 | 0 | 1
Urinary tract infection (Infections and infestations) | 8 | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 6
Cystitis (Infections and infestations) | 1 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 5 | 3 | 7
Weight decreased (Investigations) | 6 | 3 | 3
Alanine aminotransferase increased (Investigations) | 4 | 1 | 6
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 6
Gamma-glutamyltransferase increased (Investigations) | 4 | 0 | 6
Neutrophil count decreased (Investigations) | 3 | 1 | 4
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 3
White blood cell count decreased (Investigations) | 3 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 20 | 13 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 5 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 3 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 3 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 9 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 7 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 4 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 10 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 6 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 26 | 18 | 14
Headache (Nervous system disorders) | 8 | 7 | 7
Dysgeusia (Nervous system disorders) | 7 | 7 | 5
Paraesthesia (Nervous system disorders) | 5 | 5 | 7
Dizziness (Nervous system disorders) | 6 | 6 | 3
Neuropathy peripheral (Nervous system disorders) | 4 | 3 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 3
Insomnia (Psychiatric disorders) | 6 | 4 | 4
Dysuria (Renal and urinary disorders) | 2 | 3 | 4
Pollakiuria (Renal and urinary disorders) | 1 | 3 | 4
Urinary incontinence (Renal and urinary disorders) | 3 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 4 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 22 | 24
Rash (Skin and subcutaneous tissue disorders) | 11 | 4 | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 8 | 6 | 3
Nail discolouration (Skin and subcutaneous tissue disorders) | 5 | 5 | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 9 | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 3 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 2 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 3 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 5 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 3 | 1
Nail pigmentation (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Hypertension (Vascular disorders) | 6 | 5 | 2
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 1
Influenza like illness (General disorders) | 3 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 3 | 0
Hydronephrosis (Renal and urinary disorders) | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual publications will be allowed before publication of the multicenter results except as agreed with Corcept. The Investigator agrees to submit all manuscripts or abstracts to Corcept for review before submission to the publisher.

DOCUMENTS (2):
  • Study Protocol (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT03776812/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT03776812/SAP_001.pdf